CLINICAL TRIAL: NCT03733483
Title: Mechanisms for Sleep/Circadian Disruption-Induced Impairments in Bone Formation
Brief Title: Sleep Disruption Induced Impairments in Bone Formation
Acronym: SIIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-0015; K23AR070275 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Bone; Sleep Restriction

STUDY DESIGN:
Intervention Model Description: Subjects are their own controls, with baseline measurements serving as the control values prior to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Deprivation (Experimental)
  Interventions: Behavioral: Sleep Deprivation

INTERVENTIONS:
Behavioral: Sleep Deprivation — Participants in this arm will sleep for 8 hours at their habitual time for 1 week outpatient. Food will be provided for the outpatient week by the study. After the outpatient week participants will check into our inpatient Clinical Translational Research Center (CTRC) for a 9 day inpatient stay. During their inpatient stay participants will be sleep restricted to a 5 hour/night sleep opportunity for nights 2-7 of their inpatient stay. Outcome measures include a 24-hour serum draw (urine and blood) which will occur on night 1 (pre) and night 8 (post). Patients will be given a 10 + hour recovery sleep period on night 8 of their inpatient stay.

SUMMARY:
This is a small intervention study with healthy males aged 20-65 years old who habitually sleep 7-9 hours/night.This study investigates if and how sleep restriction, independent of circadian misalignment (e.g. shift work, jet lag), induces a decrease in the bone formation marker Procollagen I Intact N-Terminal Propeptide (PINP). The specific aim is to evaluate the mechanistic underpinnings for the relationship between sleep restriction and suppression of bone formation. The study will enroll 12 healthy male participants and have a two-week intervention after enrollment.

ELIGIBILITY:
Inclusion Criteria:

o Adult men aged 20-65 years old who habitually sleep 7-9 hours/night.

Exclusion Criteria:

* Regularly go to sleep after midnight;
* Shift work 1 year prior to study;
* Travel >1 time zone 4 weeks prior to study or need to travel during study;
* More than moderate activity level (>3 days of exercise per week >30 min of exercise per session);
* Current smokers (or within the previous year of study);
* Positive drug test at screening or laboratory admission;
* BMI > 30 kg/m2;
* Individuals who are concurrently participating in another research protocol that would influence their safe participation in this study. For example, participants involved in a study that requires blood draws or ingestion of experimental medication as this would increase the risk of participation in our study and/or compromise study results.
* Any clinically significant unstable medical or surgical condition within the last year (treated or untreated), including history of a clinically significant abnormality of the neurological system (including cognitive disorders or significant head injury) or any history of seizure (including febrile seizure-sleep loss has been used clinically to induce seizures in patients with epilepsy). Given the wide range of illnesses that are encountered in medical practice, it would not be possible to provide a comprehensive list of each and every disease that could serve as grounds for exclusion for the subject. However, the following is a list of illness categories that would certainly be grounds for exclusion: Connective Tissue and Joint Disorders; Neurologic/cognitive Disorders; Musculoskeletal Disorders; Immune Disorders; Chronobiologic Disorders; Cardiovascular Disorders; Respiratory Disorders; Kidney Disorders; Infectious Diseases; Hematopoietic Disorders; Neoplastic Diseases; and Endocrine and Metabolic Diseases.
* Self-reported or newly diagnosed medical condition that is still being investigated or is not under good control, including those identified on screening labs such as:

  * Out-of-range values measured on a fasting blood sample: glucose > 100 mg/dl, thyroid stimulating hormone <0.5 or >5.0 uU/ml, abnormal alkaline phosphatase <39 or >117 U/l, creatinine, or hemoglobin <14.5 g/dl men
* Any clinically significant psychiatric condition, as defined by DSM-V. Individuals with a history of most psychiatric illnesses or psychiatric disorders will be excluded, such as but not limited to depression, anxiety, alcoholism, drug dependency, schizophrenic disorders, and personality disorders (performed by medical history and physician interview). However, a personal history of limited prior counseling, psychotherapy (e.g., for adjustment reactions) will NOT be exclusionary. Evaluation of Psychiatric/Psychological Suitability:

  * Subjects must demonstrate a full understanding of the requirements and demands of the study.
  * Each subject will complete psychological screening questionnaires. Exclusionary: Center for Epidemiological Studies Depression (CES-D) ≥ 16;. Subject responses to the CES-D are reviewed immediately and appropriate referrals are made if necessary.
  * Individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressants, neuroleptic medications or major tranquilizers will be excluded from study.
  * Use of anti-depressants or any like therapeutics prescribed by a physician is exclusionary
* Individuals with any clinically significant sleep disorder; Diagnosis or symptoms of sleep disorders (history of significant parasomnia as an adult [night terrors, frequent sleep walking], insomnia, including but not limited to hypersomnias such as apnea, periodic limb movements, narcolepsy). Sleep disorders will be screened by self-report and physician interview including use of validated sleep questionnaires (PSQI, Epworth sleepiness scale, and Berlin sleep questionnaire for sleep apnea).
* Individuals on medications known to affect bone turnover (e.g. glucocorticoids, osteoporosis medications);
* Use of medications/supplements/drugs that impact sleep or bone metabolism (such as but not limited to sleep medications, marijuana etc.) within one month (participants can be studied at a later date).
* Dwelling below Denver altitude (1,600 m) 6 months prior to testing;
* Greater than moderate caffeine (>500 mg/day) or alcohol use (>14 standard drinks/week or >5 drinks in one sitting);
* Subjects with a history of heparin-induced thrombocytopenia (HIT) or an allergy to heparin;
* Inability to travel to the CU-AMC campus for study visits.
* Individuals with restrictive diets (e.g., vegan)
* Individuals with 25OHD < 20 ng/mL;
* Individuals with eGFR < 60 mL/min/1.73m2 as this is known to affect CTX measurements;
* T-score ≤ -2.5 (men ≥50 years old) or Z-score < -2.0 (men <50 years old) for bone mineral density (BMD) at the L-spine, femoral neck, or total hip on baseline DXA as compared to the DXA machine's normative database;
* Symptoms of active illness (e.g., fever); note that subject can be studied at a later date.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Swanson, MD, MCR, Principal Investigator — University of Colorado, Denver
Locations (1):
- Clinical & Translational Research Centers (CTRC) UCHealth, Aurora, Colorado, United States

REFERENCES:
- [Background] Swanson CM, Shea SA, Wolfe P, Cain SW, Munch M, Vujovic N, Czeisler CA, Buxton OM, Orwoll ES. Bone Turnover Markers After Sleep Restriction and Circadian Disruption: A Mechanism for Sleep-Related Bone Loss in Humans. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3722-3730. doi: 10.1210/jc.2017-01147. PMID 28973223
- [Derived] Swanson CM, Shanbhag P, Tussey EJ, Rynders CA, Wright KP Jr, Kohrt WM. Bone Turnover Markers After Six Nights of Insufficient Sleep and Subsequent Recovery Sleep in Healthy Men. Calcif Tissue Int. 2022 Jun;110(6):712-722. doi: 10.1007/s00223-022-00950-8. Epub 2022 Feb 8. PMID 35133471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep Deprivation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sleep Deprivation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Pro-collagen 1 Intact N-terminal Propeptide (P1NP)
Description: A marker of bone formation
Time Frame: 24 hour serum draw before and after 6 night sleep restriction. Pre measures taken on night 1 through day 2. Post measures taken on night 7 through day 8. A fasting blood sample will be taken each morning of the inpatient stay.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Sleep Deprivation
Number analyzed (Participants) | 12
ng/mL
  Baseline | 72.1 (4.4)
  Sleep Restricted | 67.4 (4.4)
Statistical Analysis 1: Comparison: Sleep Deprivation; Test type: Equivalence — Maximum likelihood estimates in a repeated measures model were used to assess the effect of insufficient sleep on P1NP levels. Change in P1NP in response to insufficient sleep was assessed using values measured every two hours on two, 24-h profiles obtained at baseline and on night 6 of sleep restriction. Circadian rhythmicity was included in the repeated-measures model as diurnal variation has been documented in prior studies. Data are presented as estimate ± standard error of the estimate; p = 0.53, Mixed Models Analysis

2. Secondary Outcome: Change in Serum C-telopeptide of Type 1 Collagen (CTX)
Description: A marker of bone resorption
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Sleep Deprivation
Number analyzed (Participants) | 12
ng/mL
  Baseline | 0.197 (0.05)
  Sleep Restricted | 0.459 (0.06)
Statistical Analysis 1: Comparison: Sleep Deprivation; Test type: Equivalence — Maximum likelihood estimates in a repeated measures model were used to assess the effect of insufficient sleep on CTX levels. Change in CTX in response to insufficient sleep was assessed using values measured every two hours on two, 24-h profiles obtained at baseline and on night 6 of sleep restriction. Circadian rhythmicity was included in the repeated-measures model as diurnal variation has been documented in prior studies. Data are presented as estimate ± standard error of the estimate; p = 0.10, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events data were collected while subjects were enrolled in the study. This included during their screening visit and during the 16 -37 days they were enrolled in the study.
Arm/Group | Sleep Deprivation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleep Deprivation (N=12)
Dry eyes (Eye disorders) | 1 (1) — One participant experienced eye discomfort during the inpatient sleep restriction portion of the study. This was resolved with saline eye drops
Irritation (Skin and subcutaneous tissue disorders) | 1 (1) — One participant experienced skin irritation due to the tape used with our IV catheter. Skin irritation resolved within 7 days.

LIMITATIONS AND CAVEATS:
1) A protocol deviation resulted in slightly longer sleep duration on one night in one participant. Results were unchanged when data were re-analyzed without data from that participant. 2) This data was from a small cohort of young, healthy, physically active men. 3) Activity restrictions imposed during sleep restriction may not accurately reflect activity during real-life sleep restriction. 4) Study diets provided may not accurately replicate real-life changes in diet due to sleep restriction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03733483/Prot_SAP_001.pdf